CLINICAL TRIAL: NCT04437381
Title: Molecular Targets for the Treatment of Histiocytosis
Acronym: TARGET-HISTIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Cancer Institute, France (Other Government); Direction de l'Hospitalisation et de l'Organisation des Soins (Unknown); Versailles Saint-Quentin-en-Yvelines University, Paris-Saclay University (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP200137
Record Dates: First submitted 2020-06-08; First posted 2020-06-18 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Histiocytosis
Keywords: histiocytosis
MeSH Terms: conditions — Histiocytosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue and blood samples and derived nucleic acids.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective: to develop technical and operating procedures for detection mutations of histiocytosis during clinical practice of no-specialized molecular platforms, for diagnosis and follow-up of the disease.

The secondary objectives: to describe therapeutic target mutations in histiocytosis patients, and to develop the cellular tests to evaluate in vitro the sensibility of these mutations drive to inhibitors.

DETAILED DESCRIPTION:
The study is ancillary of the French "Gene Histio" cohort (patients already included) and "HISTIO target 2020" cohort (patients recruited since may 2020).

The data base of the French registry of histiocytoses is held by Dr J. Donadieu, and localized in Trousseau hospital (APHP) 75012 Paris, France, where server and backup are kept.

5 teams contributes to the study with different role: Team 1 is responsible for histology diagnosis, selection of histiocyte- rich areas, extraction of nucleic acids and detection of the BRAF p.V600E mutations. This group is also responsible of the tissue and nucleic acids biobank.

Team 2 is responsible for the collection of clinical data and tissue and blood samples of the children. This group is also responsible of the clinical data base.

Team 3 is responsible for the collection of clinical data and tissue and blood samples of the adult patients.

Team 4 is responsible for the development and validation of the new methods of detection of genetic somatic alterations described in project, and will perform most of the molecular analyses and interpretations.

Team 5 is responsible for regulatory requirements preparation and submissions and takes care of replying to regulatory comments and amendments until getting approvals. The project manager will also take care of the coordination of all activities related to the database setting and utilization, liaising between researchers, doctors and operational team. Team 5 will be in charge of the data management of the database and will ensure collection tools, integration and availability of data at appropriate quality. The data manager ensures that data is collected, validated, complete, and consistent, to provide a high quality and comprehensive database to the statistics team. Team 5 includes also a statistician who will perform data analysis according to a detailed statistical analysis plan to be developed once the project is approved.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven histiocytosis;
* Informed consent form signed by patients (or parents/legal tutors of children) to participate"Gene Histio" or "HISTIO target 2020".

Exclusion Criteria:

- Patient refusal.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Paediatric and adult patients with histologically proven histiocytosis, included in either "Gene Histio" or "HISTIO target 2020" cohorts between 1997 and 2023.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Molecular alterations in histiocytosis | throughout of the study, an average of 3 years
  Characterize the molecular alterations of nucleic acids in histiocytosis. Assess the frequency and type of drugable mutations in the different sub-types and localizations of histiocytosis Molecular alterations will be assessed by next analysis of DNA or RNA extracted from histiocytosis tissue or blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François EMILE, MD, PhD, Principal Investigator — Department of Pathology, Ambroise Paré hospital, APHP
Locations (3):
- France (3):
  - Biological research center, Ambroise Paré hospital, APHP, Boulogne-Billancourt
  - Department of internal Medicine, Pitié-Salpétrière hospital, APHP, Paris
  - Department of Pediatrics, Trousseau hospital, APHP, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bigenwald C, Roos-Weil D, Pages A, Helias-Rodzewicz Z, Copie-Bergman C, Nashvi M, Khneisser P, Parrens M, Traverse-Glehen A, Ray-Coquard I, Ysebaert L, Marchand T, Razanamahery J, Charlotte F, Neel A, Damaj G, Dion J, Nazal-Traissac EM, Tardy S, Salmeron G, Monjanel H, Idbaih A, Heritier S, Haroche J, Donadieu J, Emile JF. Characterization and treatment outcomes of malignant histiocytoses in a retrospective series of 141 cases in France. Blood Adv. 2025 May 27;9(10):2530-2541. doi: 10.1182/bloodadvances.2024015208. PMID 40009752